CLINICAL TRIAL: NCT03707743
Title: A Physician-initiated, International, Multi-center, Prospective and Retrospective, Non Randomized, Observational Registry of Patients With Acute/Subacute Type B Aortic Dissection Treated by Means of the STABILISE Technique.
Brief Title: Registry of Patients With Acute/Subacute Type B Aortic Dissection Treated by Means of the STABILISE Technique (STABILISE)
Acronym: STABILISE
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Germano Melissano, MD, IRCCS San Raffaele
Other Study IDs: STABILISE
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate results of patients treated with the STABILISE technique for acute/subacute aortic dissection. Results and postoperative events are reported in accordance with the current reporting standards for endovascular aortic repair prepared and revised by the Ad Hoc Committee for Standardized Reporting Practices in Vascular Surgery of The Society for Vascular Surgery/American Association for Vascular Surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥ 18 years of age;
* Patients presenting with an acute (up to two weeks from the onset) and subacute (between 3 and 12 weeks from the onset) type B dissection with a proximal suitable non-dissected landing zone in the aortic arch or descending thoracic aorta (supra-aortic trunks debranching may be employed to obtain an adequate proximal landing zone);
* Total aortic diameter of the abdominal aorta (from supra-celiac to infra-renal level) must not exceed 42 mm;
* Patients able to sign specific informed consent for the study.

Exclusion Criteria:

* Patients with chronic type B aortic dissection (more than 12 weeks from the onset);
* Patients with acute type B aortic dissection not treated according to the following treatment protocol;
* Unwilling or unable to comply with the follow-up schedule;
* Inability or refusal to give informed consent;
* Simultaneously participating in another investigative device or drug study;
* Frank rupture;
* Systemic infection (eg, sepsis);
* Allergy to stainless steel, polyester, solder (tin, silver), polypropylene, nitinol, or gold;
* Untreatable reaction to contrast, which, in the opinion of the investigator, cannot be adequately premedicated;
* Surgical or endovascular AAA repair within 30 days before or after dissection repair;
* Previous placement of a thoracic endovascular graft;
* Prior open repair involving the descending thoracic aorta, including the supra-renal aorta and/or arch;
* Interventional and/or open surgical procedures (unrelated to dissection) within 30 days before or after dissection repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute/subacute type B aortic dissection treated by means of the STABILISE technique
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Technical success of the STABILISE procedure | 30 day
  patency of visceral vessels and iliac arteries
Clinical success | 30 day
  absence of major adverse events (mortality, neurological complications, cardiological complications, respiratory complications, intestinal ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Germano Melissano, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (34):
- United States (9):
  - Falk Cardiovascular Research Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cooper University Health Care, Camden, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Mayo Clinic, Rochester, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Knight Cardiovascular Institute, Portland, Oregon
- Australia (2):
  - Austin Hospital Heidelberg, Victoria Park, Australia
  - St Vincent's Private Hospital Melbourne, Melbourne, Victoria
- Herz Im Zentrum, Neulengbach, Hauptplatz, Austria
- Centervasc-Rio, Rio de Janeiro, Brazil, Brazil
- France (2):
  - Hopital de la Timone, Marseille, France
  - Hôpital Européen Georges Pompidou, Paris, Paris
- Germany (4):
  - Klinikum Nürnberg Süd, Nuremberg, Franconia
  - Johannes Gutenberg-University, Hamburg, Germany
  - German Aortic Center Hamburg, Hamburg, Hamburg
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
- Italy (7):
  - ASST Lecco, Lecco, Italy
  - IRCCS San Raffaele Hospital, Milan, Italy
  - AOU Modena, Modena, Italy
  - AOU Policlinico Umberto I, Roma, Italy
  - Ospedale San Giovanni di Dio, Florence
  - Ospedale Civile SS. Annunziata, Sassari
  - AOUI Verona, Verona
- Maastricht Heart+Vascular Center, Maastricht, Netherlands, Netherlands
- Waikato Hospital, Hamilton, New Zealand
- Bristish Hospital XXI / Instituto Cardiovascular de Lisboa, Lisbon, Portugal, Portugal
- Hospital Clínic de Barcelona, Barcelona, Catalonia, Spain
- University of Lund, General Hospital, Malmö, Malmo, Sweden, Sweden
- University School of Medicine Department of Cardiovascular Surgery, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Royal Brompton & Harefield NHS Foundation, Chelsea, London
  - London Guy's & St Thomas' NHS Foundation Trust, London, London

REFERENCES:
- [Background] Fattori R, Cao P, De Rango P, Czerny M, Evangelista A, Nienaber C, Rousseau H, Schepens M. Interdisciplinary expert consensus document on management of type B aortic dissection. J Am Coll Cardiol. 2013 Apr 23;61(16):1661-78. doi: 10.1016/j.jacc.2012.11.072. PMID 23500232
- [Background] Nienaber CA, Kische S, Zeller T, Rehders TC, Schneider H, Lorenzen B, Bunger C, Ince H. Provisional extension to induce complete attachment after stent-graft placement in type B aortic dissection: the PETTICOAT concept. J Endovasc Ther. 2006 Dec;13(6):738-46. doi: 10.1583/06-1923.1. PMID 17154712
- [Background] Melissano G, Bertoglio L, Rinaldi E, Civilini E, Tshomba Y, Kahlberg A, Agricola E, Chiesa R. Volume changes in aortic true and false lumen after the "PETTICOAT" procedure for type B aortic dissection. J Vasc Surg. 2012 Mar;55(3):641-51. doi: 10.1016/j.jvs.2011.10.025. Epub 2012 Jan 28. PMID 22285874
- [Background] Lombardi JV, Cambria RP, Nienaber CA, Chiesa R, Teebken O, Lee A, Mossop P, Bharadwaj P; STABLE investigators. Prospective multicenter clinical trial (STABLE) on the endovascular treatment of complicated type B aortic dissection using a composite device design. J Vasc Surg. 2012 Mar;55(3):629-640.e2. doi: 10.1016/j.jvs.2011.10.022. Epub 2011 Dec 9. PMID 22169668
- [Background] Melissano G, Bertoglio L, Rinaldi E, Mascia D, Kahlberg A, Loschi D, De Luca M, Monaco F, Chiesa R. Satisfactory short-term outcomes of the STABILISE technique for type B aortic dissection. J Vasc Surg. 2018 Oct;68(4):966-975. doi: 10.1016/j.jvs.2018.01.029. Epub 2018 Mar 30. PMID 29606568
- [Background] Hofferberth SC, Nixon IK, Boston RC, McLachlan CS, Mossop PJ. Stent-assisted balloon-induced intimal disruption and relamination in aortic dissection repair: the STABILISE concept. J Thorac Cardiovasc Surg. 2014 Apr;147(4):1240-5. doi: 10.1016/j.jtcvs.2013.03.036. Epub 2013 Apr 17. PMID 23601749
- [Background] Fillinger MF, Greenberg RK, McKinsey JF, Chaikof EL; Society for Vascular Surgery Ad Hoc Committee on TEVAR Reporting Standards. Reporting standards for thoracic endovascular aortic repair (TEVAR). J Vasc Surg. 2010 Oct;52(4):1022-33, 1033.e15. doi: 10.1016/j.jvs.2010.07.008. No abstract available. PMID 20888533
- [Background] Chaikof EL, Fillinger MF, Matsumura JS, Rutherford RB, White GH, Blankensteijn JD, Bernhard VM, Harris PL, Kent KC, May J, Veith FJ, Zarins CK. Identifying and grading factors that modify the outcome of endovascular aortic aneurysm repair. J Vasc Surg. 2002 May;35(5):1061-6. doi: 10.1067/mva.2002.123991. No abstract available. PMID 12021728
- [Background] Dake MD, Thompson M, van Sambeek M, Vermassen F, Morales JP; DEFINE Investigators. DISSECT: a new mnemonic-based approach to the categorization of aortic dissection. Eur J Vasc Endovasc Surg. 2013 Aug;46(2):175-90. doi: 10.1016/j.ejvs.2013.04.029. Epub 2013 May 28. PMID 23721817
- [Background] Riambau V, Bockler D, Brunkwall J, Cao P, Chiesa R, Coppi G, Czerny M, Fraedrich G, Haulon S, Jacobs MJ, Lachat ML, Moll FL, Setacci C, Taylor PR, Thompson M, Trimarchi S, Verhagen HJ, Verhoeven EL, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus ES, Hinchliffe RJ, Kakkos S, Koncar I, Lindholt JS, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Kolh P, Black JH 3rd, Busund R, Bjorck M, Dake M, Dick F, Eggebrecht H, Evangelista A, Grabenwoger M, Milner R, Naylor AR, Ricco JB, Rousseau H, Schmidli J. Editor's Choice - Management of Descending Thoracic Aorta Diseases: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):4-52. doi: 10.1016/j.ejvs.2016.06.005. No abstract available. PMID 28081802